CLINICAL TRIAL: NCT03035812
Title: Prospective Evaluation of Oral Alkalinization by Urologists and Nephrologists: Evolution of the Extracellular Compartment
Brief Title: Alkalinization by Urologists & Nephrologists
Acronym: AlcalUN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jean-Philippe Bertocchio (Other)
Responsible Party: Sponsor-Investigator, Jean-Philippe Bertocchio, President, Investigator, Club des Jeunes Néphrologues
Organization: Club des Jeunes Néphrologues (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AlcalUN
Record Dates: First submitted 2017-01-26; First posted 2017-01-30 (Estimated); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Metabolic Acidosis; Nephrolithiasis; Extracellular Alteration; Blood Pressure; Body Weight
Keywords: Bicarbonate
MeSH Terms: conditions — Acidosis; Nephrolithiasis; Body Weight | interventions — Alkalies; Bicarbonates; Citric Acid

STUDY DESIGN:
Intervention Model Description: Clinical and biological evaluation before and after an oral alkalinization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Alkali (Experimental): Patients in whom an oral alkalinization whatever the formulation
  Interventions: Drug: Alkali

INTERVENTIONS:
Drug: Alkali — Oral intake of alkali therapy whatever the formulation (alkali-based water, powder or pharmaceutics)
  Other Names: Bicarbonate; Citrate

SUMMARY:
Metabolic acidosis recovers a wide range of diseases in which an oral alkalinization could be useful. This therapeutic intervention has been said to increase extracellular volume leading to rising blood pressure. No prospective data has been published in clinical routine. Here, investigators propose to follow patients in which an oral alkalinization is indicated: blood pressure, body weight, and a clinical evaluation of the extracellular compartment will be performed at the beginning and during the follow-up of participants. The principal criterion of evaluation will be the variation in the extracellular compartment.

DETAILED DESCRIPTION:
Metabolic acidosis recovers a wide range of diseases - chronic kidney diseases, nephrolithiasis, or others - in which an oral alkalinization could be useful. Oral alkalinization could be performed or by bicarbonate contained in alkaline-based waters or drug therapies or by citrate. This therapeutic intervention has been said to increase extracellular volume leading to rising blood pressure, especially due to the amount of daily sodium load. No prospective data has been published in clinical routine, studying its effects on extracellular volume nor the blood pressure control.

Here, investigators propose to follow patients in which an oral alkalinization is indicated: blood pressure, body weight, and a clinical evaluation of the extracellular compartment will be performed at the beginning and during the follow-up of participants. Initial recorded data will be: age, gender, prescription (indication, kind of alkali therapy, volume and duration), body weight, body length, a clinical appreciation of the extracellular compartment, blood pressure, comorbidities, drug therapy, blood and urine composition. The recorded follow-up will be: the adherence to treatment, body weight, body length, a clinical appreciation of the extracellular compartment, blood pressure, adverse events, blood and urine composition.

The principal criterion of evaluation will be the variation in the extracellular compartment.

ELIGIBILITY:
Inclusion Criteria:

* > or = to 18 years old
* in whom an oral alkalinization is indicated

Exclusion Criteria:

* if the patient mentions its opposition to his/her enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2020-02-21 (Actual); Study Completion 2020-02-21 (Actual)

PRIMARY OUTCOMES:
Extracellular compartment M3 | At M3 (month 3)
  Evaluation of the extracellular compartment by a composite clinical outcome at M3 composed by: body weight (kg), blood pressure (in mmHg, systolic and diastolic), and the presence edema

SECONDARY OUTCOMES:
Natremia (mM) | At M3 (month 3)
  Evaluation of the impact of oral alkali therapy on natremia (mM)
Urine output (l/d) | At M3 (month 3)
  Evaluation of the impact of oral alkali therapy on urine output (l/d)
Extracellular compartment M6 | At M6 (month 6)
  Evaluation of the extracellular compartment by a composite clinical outcome at M6 composed by: body weight (kg), blood pressure (in mmHg, systolic and diastolic), and the presence edema
Kalemia (mM) | At M3 (month 3)
  Evaluation of the impact of oral alkali therapy on kalemia (mM)
Blood chloride (mM) | At M3 (month 3)
  Evaluation of the impact of oral alkali therapy on blood chloride (mM)
Bicarbonatemia (mM) | At M3 (month 3)
  Evaluation of the impact of oral alkali therapy on bicarbonatemia (mM)
Proteinemia (g/l) | At M3 (month 3)
  Evaluation of the impact of oral alkali therapy on proteinemia (mM)
Albuminemia (g/l) | At M3 (month 3)
  Evaluation of the impact of oral alkali therapy on albuminemia (mM)
Creatininemia (microM) | At M3 (month 3)
  Evaluation of the impact of oral alkali therapy on creatininemia (mM)
Natriuresis (mmol/d) | At M3 (month 3)
  Evaluation of the impact of oral alkali therapy on natriuresis (mmol/d)
Urine chloride (mmol/d) | At M3 (month 3)
  Evaluation of the impact of oral alkali therapy on urine chloride (mmol/d)
Proteinuria (g/d) | At M3 (month 3)
  Evaluation of the impact of oral alkali therapy on proteinuria (g/d)
Creatinuria (mmol/d) | At M3 (month 3)
  Evaluation of the impact of oral alkali therapy on creatinuria (mmol/d)

CONTACTS AND LOCATIONS:
Overall Officials: Julie Beaume, MD, Principal Investigator — Club des Jeunes Néphrologues
Locations (18):
- France (18):
  - Centre Hospitalier Pierre Oudot - Bourgoin-Jallieu, Bourgoin
  - La Cavale Blanche Hospital, Brest
  - CHMS Chambery, Chambéry
  - University Hospital of Grenoble, Grenoble
  - Calydial, Irigny
  - E.C.H.O. (Expansion des Centres d'Hémodialyse de l'Ouest), Le Mans
  - La Conception University Hospital, AP-HM, Marseille
  - Institut Phocéen de Néphrologie, Clinique Bouchard, Marseille
  - Uninversity Hospital of Nantes, Nantes
  - AURA Paris Plaisance, Paris
  - European Georges Pompidou Hospital, Paris
  - Tenon Hospital, AP-HP, Paris
  - Maison Blanche Hospital, Reims
  - Rennes Hospital, Rennes
  - Aub Sante, St-Malo
  - Clinic area, Strasbourg
  - Clinique Sainte Anne, Strasbourg
  - HIA Sainte-Anne, Toulon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Beaume J, Figueres L, Bobot M, de Laforcade L, Ayari H, Dolley-Hitze T, Gueutin V, Braconnier A, Golbin L, Citarda S, Seret G, Belaid L, Cohen R, Luque Y, Larceneux F, Seervai RNH, Overs C, Bertocchio JP; Club des Jeunes Nephrologues. Sodium Bicarbonate Prescription and Extracellular Volume Increase: Real-world Data Results from the AlcalUN Study. Clin Pharmacol Ther. 2022 Jan;111(1):252-262. doi: 10.1002/cpt.2427. Epub 2021 Oct 11. PMID 34564842